CLINICAL TRIAL: NCT02895737
Title: PROTECT TAVI - Prospective Randomized Outcome Study in TAVI Patients Undergoing Periprocedural Embolic Cerebral Protection With the Sentinel™ Device
Acronym: PROTECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 290/16s
Record Dates: First submitted 2016-09-06; First posted 2016-09-12 (Estimated); Last update posted 2021-03-04 (Actual); Status verified 2021-01

CONDITIONS: Cerebral Embolization During TAVI Using Balloon-expandable vs. Self-expandable Valves
Keywords: aortic stenosis, transcatheter aortic valve replacement, stroke, ischemic infarction, cerebral embolic protection device
MeSH Terms: conditions — Aortic Valve Stenosis; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (4):
- balloon-expandable TAVI without cerebral protection (Other): Patient receives a balloon-expandable transcatheter aortic valve replacement without cerebral protection
  Interventions: Device: TAVI: Edwards SAPIEN 3, Edwards Lifesciences, Edwards Sapien Ultra
- balloon-expandable TAVI with cerebral protection (Other): Patient receives a balloon-expandable transcatheter aortic valve replacement with cerebral protection
  Interventions: Device: TAVI: Edwards SAPIEN 3, Edwards Lifesciences, Edwards Sapien Ultra; Sentinel™ Cerebral Protection Systems
- self-expandable TAVI without cerebral protection (Other): Patient receives a self-expandable transcatheter aortic valve replacement without cerebral protection
  Interventions: Device: TAVI: CoreValve® Evolut R™, CoreValve Medtronic
- self-expandable TAVI with cerebral protection (Other): Patient receives a self-expandable transcatheter aortic valve replacement with cerebral protection
  Interventions: Device: TAVI: CoreValve® Evolut R™, CoreValve Medtronic; Sentinel™ Cerebral Protection Systems

INTERVENTIONS:
Device: TAVI: Edwards SAPIEN 3, Edwards Lifesciences, Edwards Sapien Ultra
  Arms: balloon-expandable TAVI without cerebral protection
Device: TAVI: Edwards SAPIEN 3, Edwards Lifesciences, Edwards Sapien Ultra; Sentinel™ Cerebral Protection Systems
  Arms: balloon-expandable TAVI with cerebral protection
Device: TAVI: CoreValve® Evolut R™, CoreValve Medtronic
  Arms: self-expandable TAVI without cerebral protection
Device: TAVI: CoreValve® Evolut R™, CoreValve Medtronic; Sentinel™ Cerebral Protection Systems
  Arms: self-expandable TAVI with cerebral protection

SUMMARY:
This prospective, randomized study was designed to analyse the difference of cerebral embolization in patients undergoing transcatheter aortic valve implantation with balloon-expandable vs. self-expandable valves by using a cerebral protection system (Sentinel™ Device).

ELIGIBILITY:
Inclusion Criteria:

* Patients with aortic stenosis and indication for transfemoral aortic valve replacement
* Freedom of significant stenosis in the area of Truncus brachiocephalicus and left A. carotis (CT)
* Necessary vessel diameter of 6.5-10 mm in the area of A. carotis communis sinistra and 9-15 mm in the area of Truncus brachiocephalicus (for delivery of protection system)
* Anomalies of aortic arch ("bovine arch" variants):

  1. Direct outflow of left A. carotis communis out of Truncus brachiocephalicus
  2. Conjoint origin of Truncus brachiocephalicus and left A. carotis communis out of aortic arch
* The patient has provided written informed consent

Exclusion Criteria:

* Apoplexy/ TIA during the last ½ year
* Severe carotid stenosis (>70%)
* Symptomatic or asymptomatic carotid stenosis with necessity of TEA or stenting
* Relevant psychiatric diseases
* Severe/ relevant visual, auditory or cognitive deficits which impede targeted anamnesis, neurologic evaluation or consenting.
* Severe neurodegenerative or progressive neuromuscular disease and state after severe craniocerebral injury with permanent neurologic sequelae and structural cerebral diseases
* Pronounced kinking/ stenosis or calcification in the area of the right A. radialis/ brachialis/ subclavia, which impede implantation of the cerebral protection system
* Significant stenosis, relevant calcifications, dissections or aneurysmatic alterations in the area of Truncus brachiocephalicus and/or A. carotis communis sinistra.
* Contraindications for MRI: among others the presence of a non-MRI-compatible pacemaker or defibrillator, metal implants in the area to be evaluated, metal fragments in the craniocerebral area, allergies, claustrophobia.
* Vessel alterations which impede among others the introduction of a 6 French sheath:

  1. Inadequate perfusion in the area of the right upper extremity (pathologic Allen´s test, vessel obstructions, peripheral vascular disease)
  2. Hemodialysis shunt, grafts, or arteriovenous fistulas in the area of right upper extremity
* Acute myocardial infarction ≤ 1 month prior to the planned procedure
* Every contraindication for the execution of a transfemoral TAVI
* Aortic annulus <19 or >29 mm
* Combined aortic vitium with predominant insufficiency.
* Severly reduced leftventricular function ≤ 20%
* Patients who are planned for a hybrid procedure (e.g. conventional operation and TAVI or simultaneous coronary intervention at coronary artery disease needing intervention) 14 days prior to the planned study procedure
* Intracardiac thrombus, hematoma, tumor or vegetations confirmed by echocardiography
* Endocarditis
* Planned concomitant procedure for atrial fibrillation (operative or via catheter ablation) during the follow up phase
* Need for emergency procedure
* Chronic drug-, medication or alcohol abuse
* Consuming disease
* Life expectancy < 1 year
* Dialysis dependency
* Patient with legal incapacity, who is not able to understand the essence, meaning and consequences of the study
* Participation in other interventional clinical trials in the month of study start or planned participation during the participation of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2016-12-28 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Total new lesion volume in protected brain regions detected by Magnetic Resonance Imaging (MRI) | Day 2-4 post-procedure

SECONDARY OUTCOMES:
Number of new cerebral lesions detected by MRI | Day 2-4 post-procedure
Occurrence of clinical stroke and/or neurocognitive dysfunction as assessed by neurological and neurocognitive assessments | Day 2-4 post-procedure; 6 months post-procedure
Postoperative Outcome according to the VARC 2 criteria | from operation until hospital discharge; 30-days, 6-months

CONTACTS AND LOCATIONS:
Locations (1):
- Deutsches Herzzentrum Muenchen, Klinik für Herz- und Gefäßchirurgie, Munich, Bavaria, Germany